CLINICAL TRIAL: NCT03669822
Title: Multi-center Acute Severe Ulcerative Colitis Cohort Study (MASCC)
Acronym: MASCC
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00174643
Record Dates: First submitted 2018-05-29; First posted 2018-09-13 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; Inflammatory bowel disease
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, stool, and colonic biopsies will be collected for a subgroup of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inpatient ulcerative colitis patients: Patients hospitalized for acute severe ulcerative colitis will be invited to enroll. Participants will be treated at the discretion of their treating physicians per standard of care. We expect some participants will be treated with standard versus accelerated infliximab dosing, permitting comparison, in addition to other treatment strategies.
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Standard of care — Care decisions driven by local physicians; this is an observational cohort.

SUMMARY:
Ulcerative colitis (UC) is a chronic, progressive immunologically mediated disease affecting nearly 1 million Americans. Up to one third of patients with UC will require hospitalization for severe disease (termed 'acute severe colitis (ASUC)'), often within the first year after diagnosis. Investigators will develop a large multi-center cohort of patients with ASUC with homogeneously collected detailed longitudinal clinical and laboratory data.

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is a chronic, progressive immunologically mediated disease affecting nearly 1 million Americans. Up to one third of patients with UC will require hospitalization for severe disease (termed 'acute severe colitis (ASUC)'), often within the first year after diagnosis. Advances in therapy for UC with the availability of effective biologics have revolutionized the medical care of UC, improving ability to achieve remission and reducing the need for colectomy for refractory disease. However, despite this general progress, investigators have not witnessed a corresponding temporal improvement in disease outcomes among those with the most severe disease. As well, providers lack the ability to 'personalize' care for UC by predicting up front which patients may develop ASUC or fail medical therapy and may benefit from early surgery, preventing protracted morbidity.

Over one-third of patients with ASUC will be refractory to intravenous steroids, the cornerstone for initial management of this condition. Infliximab and cyclosporine, the two most commonly used medical rescue therapies for this cohort, have comparable short- and long-term efficacy in two randomized controlled trials. However, up to a third of patients will not respond to such medical rescue. Lack of response is poorly understood and may be multifactorial with both patient- and drug-related factors. Among the latter, those with severe disease may have greater fecal loss of infliximab resulting in lack of efficacy. Attempts to overcome this have included accelerated induction with infliximab administered up front at a higher dose (10mg/kg) or more frequent intervals. A small single center retrospective study of only 50 patients among whom 15 received accelerated induction showed reduced short-term but not long-term rates of colectomy with this approach. However, a robust and generalizable comparison of the two infliximab induction treatment strategies are lacking. A key factor limiting study of ASUC is the lack of availability of large cohorts with detailed clinical information and linked specimens.

Here, investigators will develop a large multi-center cohort of patients with ASUC with homogeneously collected detailed longitudinal clinical and laboratory data. To the investigators' knowledge, this will be the first of its kind in the United States, and will be a key resource to understand the natural history, risk stratify and optimize therapeutic algorithms for care of patients with ASUC. A sub-study with blood, stool and biopsy specimens can be utilized for translational research into mechanisms of lack of response and development of biomarkers. The infrastructure of this network will also serve as a valuable resource for clinical trials of new therapies and novel strategies, a significant unmet need.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-80 years
* UC or IBD-unspecified (IBDU) diagnosed according to standard criteria
* Active disease defined as Simple Clinical Colitis Activity Index > 2 (day/night bowel frequency, urgency with defecation, blood in stool, general well-being, and extracolonic features)
* Admitted to the hospital
* Initiating intravenous corticosteroid therapy or medical rescue therapy

Exclusion Criteria:

* Patients with quiescent disease
* Inability to provide informed consent
* Prior colitis related surgery including J-pouch or stoma
* Non-IBD related hospital admission
* Women who are pregnant (from the specimen substudy only)
* Non - English speaking

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized ulcerative colitis patients
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2018-11-10 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Inpatient response to medical management | In-hospital (approximately 1-2 weeks)
  Response assessed by the following clinical care decisions based on binary outcomes: need for more than 1 dose of infliximab (yes=1 or no=0), switch in medical therapies (yes=1 or no=0), and need for surgery (yes=1 or no=0)

SECONDARY OUTCOMES:
Long-term response to medical management | 12 months
  Response assessed by the following clinical care decisions based on binary outcomes: need for accelerated dosing of infliximab as defined by high-dose (10mg/kg) or more than 3 doses over the first 6 weeks of therapy (yes=1 or no=0), switch in medical therapies (yes=1 or no=0), and need for surgery (yes=1 or no=0)

CONTACTS AND LOCATIONS:
Locations (1):
- Joanna Melia, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided